CLINICAL TRIAL: NCT00005921
Title: An Open, Serial-Panel, Multiple-Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of L-743,872 in Patients With Candida Esophagitis
Brief Title: A Study of the Side Effects of L-743,872 in Men With Candidal Esophagitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 267A; 007-00
Record Dates: First submitted 2000-06-19; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-06

CONDITIONS: Candidiasis, Esophageal; HIV Infections
Keywords: Dose-Response Relationship, Drug; Antifungal Agents; Candidiasis; Esophageal Diseases; MK 0991
MeSH Terms: conditions — Candidiasis; HIV Infections; Esophageal Diseases | interventions — Caspofungin

INTERVENTIONS:
Drug: L-743,872

SUMMARY:
The purpose of this study is to see if it is safe to give L-743,872 to men with candidal esophagitis, an AIDS-related yeast infection in the esophagus.

DETAILED DESCRIPTION:
In this open-label study, patients receive intravenous L-743,872 every 24 hours at one of three dose levels for 14 days. Post-study safety evaluations continue for 4 weeks after the final dose. Pharmacokinetics and safety measurements are taken throughout the 6-week study.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are an 18- to 65-year-old man with candidal esophagitis.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18

CONTACTS AND LOCATIONS:
Locations (1):
- Gary Calandra, Rahway, New Jersey, United States